CLINICAL TRIAL: NCT02266680
Title: A Randomized Controlled Trial of the Effectiveness of Breathing Focused Yoga (BFY) in Improving Symptoms of Social Anxiety Disorder
Brief Title: Breathing Focused Yoga in Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Arun Ravindran, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150/2011
Record Dates: First submitted 2014-10-07; First posted 2014-10-17 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2016-09

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety; Yoga
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga Treatment Group (Experimental): BFY will be taught by a trained yoga instructor. Group sessions will be offered twice a week for 60 minutes each (i.e., a total of 2 hours per week), for 8 weeks.
  Interventions: Behavioral: Yoga Treatment Group
- Waitlist Group (No Intervention): Waitlisted participants will receive BFY at the next available group after their waitlist period is completed

INTERVENTIONS:
Behavioral: Yoga Treatment Group — The breathing focused yoga intervention is a manualized yoga protocol developed at CAMH by the Mood and Anxiety Disorders group, with yoga teacher, Ms. Tiffany Garfinkel, as the lead. BFY incorporates postures and meditation, but there is a special focus on controlled breathing at different rates, including Ujjaji or slow inhalation, exhalation and holding of breath; Bhastrika or Kapalabhati, two types of vigorous breathing with forced exhalation; and cyclical breathing or a repeated pattern of slow, moderate and fast breathing.
  Other Names: Breathing Focused Yoga
  Arms: Yoga Treatment Group

SUMMARY:
The goal of this study is to determine the safety and effectiveness of Breathing Focused Yoga (BFY) in improving symptoms of social anxiety disorder (SAD). Patients with SAD will be randomized to 8 weeks of yoga or 8 weeks of wait-list. Symptom severity and quality of life will be compared between the two groups before and after the 8 weeks.

DETAILED DESCRIPTION:
This is an exploratory 8-week study with a randomized controlled, parallel group design, and will be carried out in two phases: 1) 8-week treatment phase and 2) a 3-month follow-up phase.

60 patients meeting Diagnostic and Statistical Manual IV Text Revision, (DSM-IV-TR), diagnostic criteria for social anxiety disorder will be recruited. Patients who have provided written consent, have met study criteria, and are stabilized on pharmacotherapy will be enrolled into the study.

In the treatment phase, patients will be randomized, to one of two groups 1) Breathing Focused Yoga (BFY); or 2) wait-list group.

A sub-set of 15 drug- naïve patients and matched healthy controls will undergo functional magnetic resonance imaging (fMRI) scans before and after yoga treatment.

A blood sample for genetic analysis will be taken from all SAD patients, to investigate to presence of genes linked to SAD and t treatment response.

The primary aim of the study is to determine the safety and effectiveness of Breathing Focused Yoga (BFY) in improving symptoms of SAD.

There are two secondary aims:

1. To enhance the limited research data on the effect of treatment on neural circuitry in SAD, the investigators will also conduct fMRI scans on SAD patients and matched healthy controls pre- and post-BFY intervention.
2. As well, to add to the literature on the genetics of SAD, the investigators will validate the links between specific gene polymorphisms and SAD that are already identified in the literature, and evaluate if they predict treatment response following BFY intervention.

Primary Hypotheses

1. Subjects with Social Anxiety Disorder will show significant improvement in symptoms after BFY, compared to the wait-list group.
2. Improvement in quality of life scores will be significantly greater in the BFY group compared to the wait-list group.

Secondary Hypotheses

1. At baseline, the fMRI indications of neural circuitry of SAD subjects will differ from that of healthy controls.
2. After yoga treatment, the fMRI indications of neural circuitry of treatment responders in the SAD group will be similar to that of healthy controls.
3. The presence of specific gene polymorphisms in SAD patients will predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-65 years
2. Primary diagnosis of SAD, per the DSM-IV-TR (APA, 2000)
3. LSAS score of ≥50
4. Absence of serious medical illness
5. Not on any psychotropic medications currently, or on stable medications for at least 8 weeks prior to starting treatment
6. Short-acting benzodiazepines (e.g. lorazepam 1 mg prn) and sleep medications (e.g. zopiclone 7.5 mg prn) may be used, but not within 12 hours prior to a study visit

Exclusion Criteria:

1. Current primary diagnosis of major depressive episode, mania or psychosis
2. A score of ≥15 on the first 17 items of the HAM-D at Screening or Baseline
3. Diagnosis of a substance abuse disorder within the prior 6 months
4. Presence of medical or mental health conditions that would inhibit the patient's ability to participate in the study
5. Currently receiving any structured formal psychotherapy (supportive therapy is allowed)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Liebowitz Social Anxiety Scale (LSAS) Total Score | Baseline to study endpoint (Week 8)

SECONDARY OUTCOMES:
Change in Clinical Global Impression Scale | Baseline to study endpoint (Week 8)
Change in Hamilton Depression Rating Scale (HAM-D) Total Score | Baseline to study endpoint (Week 8)
Change in Quality of Life Enjoyment and Satisfaction Scale (QLESQ) Total Score | Baseline to study endpoint (Week 8)
Change in Quick Inventory of Depressive Symptomatology (QIDS) Total Score | Baseline to study endpoint (Week 8)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Ravindran, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addition and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research